CLINICAL TRIAL: NCT05421195
Title: Clinical Treatment Research of COVID-19-related Olfactory Dysfunction: A Randomized Controlled Trial
Brief Title: Clinical Treatment Research of COVID-19-related Olfactory Dysfunction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Eye & ENT Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PIOD2022-5V1
Record Dates: First submitted 2022-06-14; First posted 2022-06-16 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: Olfactory Dysfunction
Keywords: olfactory dysfunction
MeSH Terms: interventions — Olfactory Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Glucocorticoid therapy with olfactory training (Experimental): olfactory training plus oral Glucocorticoid
  Interventions: Drug: corticosteroids therapy; Other: Olfactory training
- Olfactory training (Other): Olfactory training only
  Interventions: Other: Olfactory training

INTERVENTIONS:
Drug: corticosteroids therapy — Oral corticosteroids
  Arms: Glucocorticoid therapy with olfactory training
Other: Olfactory training — repeat and deliberate sniffing of a set of odorants

SUMMARY:
Studies have demonstrated that patients with COVID-19- related olfactory dysfunction could improve the olfactory function after olfactory training. But the efficacy of oral corticosteroids is controversial. Some evidences shown that corticosteroid treatment would benefit post-COVID-19 olfactory dysfunction and the purpose of this study is to evaluate its efficacy.

DETAILED DESCRIPTION:
Reports of COVID-19-related olfactory dysfunction describe a sudden onset of olfactory impairment, which may be in the presence or absence of other symptoms. The possibility that olfactory dysfunction could act as a marker for disease. When COVID-19-related olfactory dysfunction improves spontaneously, specific treatment may not be required. However,when impairment persists beyond 2 weeks, it may be reasonable for treatment to be considered. The efficacy of available treatments for patients with COVID-19-related olfactory dysfunction is unknown. Olfactory training involves repeat and deliberate sniffing of a set of odorants (commonly lemon, rose, cloves, and eucalyptus) for 20 seconds each at least twice a day for at least 3 months (or longer if possible). Studies have demonstrated improved olfaction in patients after olfactory training. Olfactory training can be considered for patients with persistent COVID-19-related olfactory dysfunction. Some evidences shown that corticosteroid treatment would benefit post-COVID-19 olfactory dysfunction but the evidences is not adequate. Until now, the efficacy of oral corticosteroids is controversial. This study investigate the efficacy and the safety of oral corticosteroids and olfactory training as a treatment for patients with COVID-19-related olfactory dysfunction.

ELIGIBILITY:
Inclusion Criteria:

1. Previous diagnosis of COVID-19 infection; 2. Olfactory function was normal in the past, and the olfactory function decreased due to COVID-19 infection, which has occurred more than 2 weeks; 3. Olfactory function test score: TDI ≤ 30; 4.18 ≤ age ≤ 55 years old; 5.Good overall physical condition, without other diseases that may affect the test; 6. No active infection, such as uncontrolled pneumonia; 7. Women with reproductive potential and sexually active men agree to use acceptable and effective contraceptive methods.

Exclusion Criteria:

1. Participants who refuse to sign informed consent; 2. Participants who have other diseases that affect the result, such as trauma, benign and malignant tumors of nasal cavity and paranasal sinuses, intracranial benign and malignant tumors, etc; 3. Participants with uncontrolled concurrent diseases that the researcher believes will interfere with the treatment; 4. Participants who has contraindications to oral corticosteroids, such as serious gastric and duodenal ulcer, diabetes, glaucoma, etc; 5. Participants who have serious neurological or mental diseases, including dementia and seizures; 6.Participants who have oral corticosteroids history within 2 weeks, or who have recently taken a large amount of oral corticosteroids and are not suitable after the evaluation of the researcher; 7. Participants who have used corticosteroids therapy during the treatment of COVID-19 and olfactory function didn't recover; 8. Pregnant or lactating women; 9. persons without personal freedom and independent civil capacity; 10. Participants who have been enrolled in other intervention clinical trials; 11. Participants who with autoimmune diseases; 12. Participants who has any situation that may hinder the compliance of the protocol study or the safety during the study; 13. Other situations that the investigators think are not suitable for the trial.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 124 (Estimated)
Dates: Start 2022-06-17 (Estimated); Primary Completion 2023-02-01 (Estimated); Study Completion 2023-03-01 (Estimated)

PRIMARY OUTCOMES:
Olfactory function test result：the sum of the scores of odor threshold (T), odor discrimination (D), and odor identification (I) is TDI. | 3 months
  Olfactory tests combination of odor threshold (T), odor discrimination (D), and odor identification (I). The minimum values is zero, the maximum values of odor threshold (T), discrimination (D), and identification (I) is 16, the sum of the scores is TDI, which is between 0 to 48, the higher scores mean a better outcome.

SECONDARY OUTCOMES:
Odor threshold (T), Odor Discrimination (D), Odor Identification (I) | 3 months
  The scale of odor threshold (T), discrimination (D), and identification (I).The minimum values is zero, the maximum values of odor threshold (T), discrimination (D), and identification (I) is 16, the higher scores mean a better outcome.
the Visual Analogue Scale（VAS）of olfactory function | 3 months
  Participants should value their olfactory function by use the Visual Analogue Scale（VAS), the minimum values is 0, the maximum values is 10, the higher scores mean a better outcome.
Questionnaire of Olfactory Disorders | 3 months
  every patients should answer the Questionnaire of Olfactory Disorders and record the results

CONTACTS AND LOCATIONS:
Overall Officials: Hongmeng Yu, Dr, Principal Investigator — Eye & ENT Hospital, Fudan University; Xicai Sun, Dr, Principal Investigator — Eye&ENT Hospital,Fudan University
Locations (1):
- Eye & ENT Hospital, Shanghai, Shanghai Municipality, China